CLINICAL TRIAL: NCT05746793
Title: At High-risk for Pre-eclampsia After Assisted Reproductive Technology
Acronym: HEART
Status: Recruiting | Type: Observational
Sponsor: CRG UZ Brussel (Other)
Responsible Party: Principal Investigator, Mackens Shari, Prof. Dr., CRG UZ Brussel
Other Study IDs: 22271HEART
Record Dates: First submitted 2022-11-07; First posted 2023-02-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Urine Specimen Collection; Blood Pressure Determination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — endometrial biopsy; menstrual blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subfertile polycystic ovarian syndrome (PCOS) patients undergoing ART treatment: Peripheral blood collection. MOCK frozen embryo preparative cycle. Endometrial pipelle biopsy. Collection of menstrual blood. Questionnaire. Nutritional/metabolic evaluation. Cardiac work-up. Preconceptional and prenatal ultrasound. Blood pressure measurements. Urine analysis.
  Interventions: Procedure: endometrium biopsy; Diagnostic Test: Transabdominal ultrasound; Diagnostic Test: Peripheral phlebotomy; Diagnostic Test: Urine collection; Other: MOCK frozen embryo transfer preparative cycle.; Diagnostic Test: Baseline questionnaire; Other: collection of menstrual blood; Diagnostic Test: nutritional and metabolic work-up; Diagnostic Test: cardiac work-up; Diagnostic Test: Blood pressure measurement
- Oocyte acceptors: Peripheral blood collection. MOCK frozen embryo preparative cycle. Endometrial pipelle biopsy. Collection of menstrual blood. Questionnaire. Nutritional/metabolic evaluation. Cardiac work-up. Preconceptional and prenatal ultrasound. Blood pressure measurements. Urine analysis.
  Interventions: Procedure: endometrium biopsy; Diagnostic Test: Transabdominal ultrasound; Diagnostic Test: Peripheral phlebotomy; Diagnostic Test: Urine collection; Other: MOCK frozen embryo transfer preparative cycle.; Diagnostic Test: Baseline questionnaire; Other: collection of menstrual blood; Diagnostic Test: nutritional and metabolic work-up; Diagnostic Test: cardiac work-up; Diagnostic Test: Blood pressure measurement

INTERVENTIONS:
Procedure: endometrium biopsy — The procedure is performed without any anesthesia and takes approximately 5 minutes.
  A small plastic pipelle is put through the cervix into the uterine cavity. The endometrial tissue is aspirated into the pipelle.
Diagnostic Test: Transabdominal ultrasound — Evaluation of fetal biometry and doppler flow study using ultrasound.
Diagnostic Test: Peripheral phlebotomy — single puncture collection of peripheral venous blood.
Diagnostic Test: Urine collection — Collection of urine in a plastic cup.
Other: MOCK frozen embryo transfer preparative cycle. — Start with daily estradiol (progynova, oestrogel) administration at hormonal baseline (day 2 of the cycle or with confirmation using endocrine evaluation). When adequate thickness (≥6.5 mm) of the endometrium is achieved (usually after 10-14 days), progesterone is administered daily. 6 days after progesterone administration, the pipelle biopsy will be performed. When this test cycle has ended and menstruation starts, patients will be asked to collect their menstrual flow, during the first night of heavy/red flow, in a menstrual cup. The next day patients will be asked to bring their collected menstrual blood to our center and they will undergo a blood analysis needed for the start of their ART treatment.
Diagnostic Test: Baseline questionnaire — questionnaire the patient has to fill in
Other: collection of menstrual blood — collection of menstrual blood during the first day of heavy menstrual flow for at least 6 hours
Diagnostic Test: nutritional and metabolic work-up — Including body composition analysis by BIA/whole body MRI and analysis of resting energy expenditure (REE).
Diagnostic Test: cardiac work-up — Using transthoracic ultrasound.
Diagnostic Test: Blood pressure measurement — Blood pressure measurement

SUMMARY:
The overarching goal of the project is to unravel PE etiopathogenesis in high-risk patients (PCOS patients and oocyte acceptors) after assisted reproductive technology (ART) to individualize prenatal care following ART and to determine potential targets for new PE prevention options decreasing the morbidity/mortality caused by this pathology. More specifically, the following objectives/work packages (WPs) are put forward:

* WP1 - PRECONCEPTION: Identify preconceptional maternal characteristics associated with in-creased risk of PE in ART patients (1a) and investigate the potential role of the endometrium prior to pregnancy (1b).
* WP2 - DURING PREGNANCY: Evaluate the Fetal Medicine Foundation's (FMF) first trimester PE screening in selected high-risk groups post ART to explore the clinical benefit in this specific context (2a) and investigate the association between parameters during the pregnancy and PE development post-ART.
* WP3 - AT DELIVERY: Identifying placental molecular pathways associated with PE post-ART.

DETAILED DESCRIPTION:
Background:

Pre-eclampsia (PE) is a multisystemic syndrome occurring in 4-5% of pregnant women. It is defined by a new-onset hypertension (HT) developing after 20 weeks of gestation in combination with one of the following entities: proteinuria, maternal organ dysfunction and/or uteroplacental insufficiency. The vicious circle of the syndrome can end up in life-threatening complications for mother and child and, today, the only treatment of cure is the induction of delivery. Furthermore, besides the problems in the acute phase of the disease, women who experienced PE have been shown to have an increased lifetime risk of developing cardiovascular disease (CVD) and chronic kidney disease, while the children carry the consequences of their prematurity and, often following intra-uterine growth restriction, also seem to be more prone to develop metabolic disturbances like diabetes, HT and CVD later in life. Research, including data publishes by my own research group, shows that the risk of PE development in subfertile patients undergoing assisted reproductive technology (ART), is more than doubled, with incidences between 8-12%.

ART includes in vitro fertilization (IVF) and intracytoplasmic sperm injection (ICSI), using autologous or heterologous gametes, followed by fresh or frozen embryo transfer. The increased risk of PE within this population has mainly been attributed to known maternal PE risk factors associated with ART like increased maternal age, nulliparity and metabolic disturbances e.g. in patients with polycystic ovary syndrome (PCOS). Recent studies however have shown that ART is an independent risk factor of PE. More specifically, a higher PE incidence is consistently observed when patients have a frozen embryo transfer (FET) in an artificially prepared cycle. Unlike in a natural cycle in which ovulation occurs, an artificial cycle is characterized by the absence of ovulation as the luteal phase is induced by exogenous progesterone administration. It has been put forward that the absence of the corpus luteum, producing vasoactive and angiogenic substances (e.g. VEG-F, relaxin) and thereby orchestrating a correct placental development, could be held responsible for this observation. Other high risk ART patients are recipients of heterologous oocytes (i.e. oocyte recipients) potentially due to immunological conflicts.

In 2016, the ASPRE trial published their results evaluating a new first trimester screening tool developed by the fetal medicine foundation (FMF). This algorithm takes into account a limited number of anamnestic maternal characteristics, maternal blood pressure, the measurement of placental growth factor (PlGF) as a serum biomarker and the ultrasonographic measurement of the pulsatility index of the uterine artery. When an increased risk of PE had been detected (>1/100), aspirin daily is given, starting before 16 weeks' of gestation.

As of May 2021, the FMF first trimester screening for PE is offered in the Brussels IVF fertility clinic to all the above-described high-risk patients pregnant following ART (PCOS and oocyte recipients included). Preliminary data confirm a high incidence of positive screening with an overall risk of 18%, reaching upto 27% in oocyte recipients (compared to the reported 10% in the general population following spontaneous conception). To the best of our knowledge, the applicability of the screening tool and aspirin administration for PE prevention has never been specifically evaluated post-ART. PE etiopathogenesis is complex and the exact molecular causative processes are still being unraveled. PE has a wide range of clinical presentations and it is currently unknown what drives these differences. Of critical importance for instance is the difference between early onset pre-eclampsia (EOPE), defined as PE occurring before 34 weeks of gestation and late onset pre-eclampsia (LOPE), defined as PE occurring at or after 34 weeks of gestation. In EOPE, which is mainly a placental disease, the impaired invasion of the spiral arteries by the extravillous cytotrofoblast cells has been put forward as the key pathophysiological component. This in contrary to LOPE, which is seen as a maternal disease, where there is a discrepancy between fetal growth, aging of the placenta an the maternal supply and cardiovascular reserve. Further, single-cell RNA sequencing on placentas confirmed the extensive different expressed genes between EOPE and LOPE. Also, the role of different serum markers (PlGF, sFLT-1, VEGF, leptin, annexin…) have been studied, but their contribution to EOPE and LOPE still remains unclear.

Lastly, very limited but intriguing research data suggest that the preconceptional endometrium could be implicated in PE development during pregnancy, with the focus on impaired decidualization and its role in PE origin. Given the differences in patient characteristics between the above-mentioned ART subgroups at risk for PE, our research team expects their PE-etiopathogenesis to be diverse. Though the multidisciplinary approach of this project, both on a clinical and fundamental research level, we hope to unravel pre-eclampsia, a multifactorial disease, and this in specific relation to different ART high-risk groups. This way, ultimately, the results will point towards targets for prevention and treatment of PE following ART and will contribute to a decrease in the morbidity and mortality associated with this devastating disease, for which, currently, no cure but termination of the pregnancy is available.

Hypothesis:

Work package 1a: there is a significant difference in preconceptional maternal characteristics between ART patients screening positive/developing PE and ART patients screening negative/not developing PE and these identified risk factors are specific for each ART subgroup.

Work package 1b: preconceptionally harvested endometrial tissue/stromal cells/organoids harbor significant differences in function of the subsequent (i.e. during pregnancy) negative or positive PE screening, PE development and specific high-risk ART group.

Work package 2a: the incidence of a positive screening/PE development (EOPE vs. LOPE) differs significantly among different ART groups.

Work package 2b: parameters during the pregnancy (blood pressure, biomarkers in the blood, ultrasound, nutritional and cardiac parameters) are significantly different between ART patients screening positive/developing PE and these identified parameters are specific for each ART subgroup.

Work package 3: placental tissue, membranes, cord tissue and cord blood harbor significant differences in expressed molecular pathways depending on negative or positive PE screening, PE development or not and are specific for the high-risk ART group.

Experimental design:

Prospective interventional cohort study without the use of a product nor medical device.

Methodology:

The study population will be subdivided into two different patient groups. Patients will be asked to participate to the study when they are planning to undergo ART and are (already prior to the start of their treatment) suspected to be at higher risk for the development PE after achieving pregnancy:

* Group 1 will include oocyte recipients as the use of donor oocytes predisposes them to a potential immunological conflict during pregnancy contributing to PE development
* Group 2 will include PCOS patients as endocrine and metabolic abnormalities predispose them to an abnormal trophoblast invasion contributing to PE development Work package 1a: evaluation of maternal baseline characteristics, laboratory studies, ultrasound examination, cardiac and nutritional work-up.

Work package 1b: harvesting and biobanking of preconceptional endometrium during the luteal phase of a preparative non-conceptional test-ART cycle (MOCK cycle). Depending on the outcome of the pregnancy, tissue can be thawed and used for basic research experiments (stromal cell lines, organoids, decidualization experiments, implantation experiments).

Work package 2a: patients are screened between 11- and 14-weeks' gestation using the FMF PE screening algorithm (routine care at our center). When patients are determined to be at high-risk of PE development (>1/100), they are advised to take aspirin (160 mg daily) until 36 weeks' gestation.

Work package 2b: patients will be followed up at different time points during their pregnancy (7, 12, 20, 28, 36 weeks' gestation) using urine sampling, blood analysis, blood pressure measurement, cardiac and nutritional work-up and ultrasound evaluation.

Work package 3: collection of placental tissue, membranes, umbilical cord tissue and cord blood at time of delivery for basic research analysis. Evaluation of different molecular pathways and expressed genes between no PE, EOPE and LOPE and this in specific relation to the different high-risk groups.

ELIGIBILITY:
Inclusion Criteria:

* First time oocyte acceptors Or Nulliparous PCOS patients undergoing ART (IVF/ICSI)
* Criteria for PCOS: two out of the three following criteria must be present:

  1. Oligo-or anovulation: a menstrual cycle >35 days
  2. Hyperandrogenism:

     * Clinically: the presence of hirsutism and/ or severe acne in combination with alopecia confirmed hyperandrogenism Or
     * Biochemically: serum total testosterone >52 ng/dl or calculated free testosterone >0,64 ng/dl
  3. Polycystic ovaries:

     * Follicle number per ovary (FNPO) ≥ 12 on both ovaries Or
     * Ovarian volume ≥ 10 ml in both ovaries Or
     * One ovary with ≥ 20 follicles (Using endovaginal US transducers with a frequency bandwidth that includes 8 MHz) Or
     * AMH ≥ 4,9 ng/ml

Exclusion Criteria:

* Known essential hypertension or development of a new-onset hypertension before 20 weeks' gestation

  * Hypertension is defined as a systolic blood pressure ≥ 140 or a diastolic blood pressure ≥ 90 on two separate measurements with at least 20 minutes in between, taken when the patients is in a seated position Or
  * The patient is known with hypertension, diagnosed by a certified doctor
* Known diabetes type 1 or 2 before pregnancy

  * Diagnosis of diabetes is confirmed when one of the following is present:

    * Fasting glucose ≥ 126 mg/dl
    * A 2-hour plasma glucose level ≥ 200 mg/dL during a 75-g oral glucose tolerance test Or
  * The patient is known with diabetes (type 1 or 2), diagnosed by a certified doctor
* Thyroid dysfunction not under control with medication:

  * Hyperthyroidism, the diagnoses is made when:
* Peripheral blood TSH <0,5 mIU/L and fT4 >1,9 ng/dl Or
* When the patient is known with hyperthyroidism diagnosed by a certified physician

  * Hypothyroidism, the diagnosis is made when:

    * Peripheral blood TSH >5 mIU/L and fT4 <0,7 ng/dl Or
    * When the patient is known with hypothyroidism diagnosed by a certified physician
* Other endocrinological disorder (including Cushing syndrome, Adrenal insufficiency, acromegaly): for diagnosis we will trust the opinion of the certified endocrinologist
* Cardiovascular diseases (including coronary artery disease, arrhythmia, heart valve disease and heart failure): for diagnosis we will trust the opinion of the certified cardiologist
* Renal disease/insufficiency: for diagnosis we will trust the opinion of the certified nephrologist
* Systemic lupus erythematosus: for diagnosis we will trust the opinion of the certified internal medicine doctor
* Antiphospholipid syndrome: for diagnosis we will trust the opinion of the certified internal medicine doctor
* Liver dysfunction/disease: for diagnosis we will trust the opinion of the certified gastroenterologist
* History of prior pre-eclampsia
* Women pregnant with a fetus with known abnormalities such chromosomal anomalies, structural deformities of limbs or organs or any other prebirth diagnosed syndromes or defects
* Multiple pregnancy

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patients with a womb, who want to get pregnant and present themselves at our fertility clinic.
Study Population: Patients at high-risk of developing PE and planned to undergo ART:
  * Oocyte recipients: patients are planned to undergo a transfer of an embryo conceived with a donor oocyte
  * PCOS patients: patients diagnosed with polycystic ovary syndrome (Rotterdam criteria) and planned to undergo a IVF/ICSI or IVM treatment
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
BMI (kg/m2) | 1 year
  measurement of height en weight. Work package 1: preconceptional, metabolic analysis Work package 2: during pregnancy, metabolic analysis
Total energy expenditure (kcal/day) | 1 year
  Work package 1: preconceptional, metabolic analysis Work package 2: during pregnancy, metabolic analysis
number of laps of 6MWT (number) | 1 year
  6 minute walking test Work package 1: preconceptional, metabolic analysis Work package 2: during pregnancy, metabolic analysis
Saturation beginning and end of 6MWT (%) | 1 year
  6 minute walking test Work package 1: preconceptional, metabolic analysis Work package 2: during pregnancy, metabolic analysis
pulse beginning and end of 6MWT | 1 year
  6 minute walking test Work package 1: preconceptional, metabolic analysis Work package 2: during pregnancy, metabolic analysis
Effective maximal handgrip strength (KPa) | 1 year
  Hangrip strenght Work package 1: preconceptional, metabolic analysis Work package 2: during pregnancy, metabolic analysis
Time until 50% of effective handgrip strenght (s) | 1 year
  Hangrip strenght Work package 1: preconceptional, metabolic analysis Work package 2: during pregnancy, metabolic analysis
IVSd (mm) | 1 year
  Transthoracic ultrasound Evaluation of left ventricle and left ventricle systolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
PWTd (mm) | 1 year
  Transthoracic ultrasound Evaluation of left ventricle and left ventricle systolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
LVEDD (mm) | 1 year
  Transthoracic ultrasound Evaluation of left ventricle and left ventricle systolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
IVSs (mm) | 1 year
  Transthoracic ultrasound Evaluation of left ventricle and left ventricle systolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
PWTs (mm) | 1 year
  Transthoracic ultrasound Evaluation of left ventricle and left ventricle systolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
LVESD (mm) | 1 year
  Transthoracic ultrasound Evaluation of left ventricle and left ventricle systolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
LV mass (indexed) mg/m2 | 1 year
  Transthoracic ultrasound Evaluation of left ventricle and left ventricle systolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
LVEF (visual, manual modified Simpson's biplane, auto-EF) (%) | 1 year
  Transthoracic ultrasound Evaluation of left ventricle and left ventricle systolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
LV GLS (LV MW) (-%) | 1 year
  Transthoracic ultrasound Evaluation of left ventricle and left ventricle systolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
E-wave velocity (cm/s) | 1 year
  Transthoracic ultrasound Evaluation of left ventricle diastolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
A-wave velocity (cm/s) | 1 year
  Transthoracic ultrasound Evaluation of left ventricle diastolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
Deceleration time (ms) | 1 year
  Transthoracic ultrasound Evaluation of left ventricle diastolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
E/A ratio | 1 year
  Transthoracic ultrasound Evaluation of left ventricle diastolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
Septal wall e' (cm/s) | 1 year
  Transthoracic ultrasound Evaluation of left ventricle diastolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
Lateral wall e' (cm/s) | 1 year
  Transthoracic ultrasound Evaluation of left ventricle diastolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
E/e' ratio | 1 year
  Transthoracic ultrasound Evaluation of left ventricle diastolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
Septal e'/lateral e' ratio | 1 year
  Transthoracic ultrasound Evaluation of left ventricle diastolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
LA AP diameters (mm) | 1 year
  Transthoracic ultrasound Evaluation of left atrium Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
LAESVi (mL/M2) | 1 year
  Transthoracic ultrasound Evaluation of left atrium Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
La strain (-%) | 1 year
  Transthoracic ultrasound Evaluation of left atrium Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
TAPSE (mm) | 1 year
  Transthoracic ultrasound Evaluation of right ventricle and RV systolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
RV s' (cm) | 1 year
  Transthoracic ultrasound Evaluation of right ventricle and RV systolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
RV GLS (RV MW) (-%) | 1 year
  Transthoracic ultrasound Evaluation of right ventricle and RV systolic function Work package 1: preconceptional, Work package 2: during pregnancy, cardiac evaluation
systolic, diastolic bloodpressure and mean arterial pressure (mmHg) | 1 year
  Blood pressure measurement device. Work package 1: preconception Work package 2: during pregnancy
Pulsatility index of the uterine artery | 1 year
  ultrasound Work package 1: preconception Work package 2: during pregnancy
(sub)endometrial flow (1,2,3) | 1 year
  ultrasound Work package 1: preconception Work package 2: during pregnancy
PRL mRNA expression | 3 months
  RNA sequencing Work package 1: preconception
PRL production (ng/ml) | 3 months
  ELISA Work package 1: preconception
IGFBP1 mRNA expression | 3 months
  RNA sequencing Endometrial tissue Work package 1: preconception
IGFBP1 (pg/ml) | 3 months
  ELISA Endometrial tissue Work package 1: preconception
PlGF (pg/ml) | 3 months
  blood sample Work package 1: preconception Work package 2: during pregnancy
sFLT1 (pg/ml) | 3 months
  blood sample Work package 1: preconception Work package 2: during pregnancy
sENG (ng/ml) | 3 months
  blood sample Work package 1: preconception Work package 2: during pregnancy
Incidence of positive PE screening (%) | 6 months
  Fetal medicine foundation screening algorithm. Work package 2: during pregnancy
Estimated fetal weight (g) | 1 year
  ultrasound Work package 2: during pregnancy
PI umbilical artery | 1 year
  ultrasound Work package 2: during pregnancy
PI uterine artery | 1 year
  ultrasound Work package 2: during pregnancy
gestational age at diagnoses PE (weeks) | 1 year
  work package 2: during pregnancy
incidence of PE (%) | 1 year
  work package 2: during pregnancy
severity of PE (mild/severe) | 1 year
  work package 2: during pregnancy
gestational age at delivery (weeks) | 1 year
  work package 3: at delivery
birth weight (grams) | 1 year
  work package 3: at delivery
APGAR scores of baby after 1, 5 and 10 minutes (1-10) | 1 year
  work package 3: at delivery
different expressed genes (DEGs) of placenta's | 1 year
  work package 3: at delivery RNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Shari Mackens, PhD, MD, Principal Investigator — Medical director Brussels IVF
Locations (1):
- Brussels IVF, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided